CLINICAL TRIAL: NCT01920620
Title: Inpatient Obesity: Can Weight Loss Intervention During Hospitalization Lead to Sustained Weight Loss at Six Months Following Discharge?
Brief Title: Inpatient Obesity Intervention With Phone Follow-up
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Kelley Wachsberg, Assistant Professor, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Obesity Intervention NU
Record Dates: First submitted 2013-08-08; First posted 2013-08-12 (Estimated); Last update posted 2016-01-20 (Estimated); Status verified 2016-01

CONDITIONS: Obesity
Keywords: obesity, inpatient, intervention, weight loss
MeSH Terms: conditions — Obesity; Weight Loss | interventions — Motivational Interviewing

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention Arm (Experimental): Inpatient weight loss counseling Motivational interviewing and troubleshooting via phone
  Interventions: Behavioral: Inpatient weight loss counseling; Behavioral: Motivational interviewing and troubleshooting via phone
- Usual Care Arm (No Intervention): Participants in the usual care group were not provided with any specific instructions regarding weight loss, diet or exercise prior to discharge. Follow-up phone calls for usual care subject were used only to obtain weight and assess for changes in medications or health condition.

INTERVENTIONS:
Behavioral: Inpatient weight loss counseling — Weight loss counseling utilizing a 13 minute patient education video on weight loss and an 25 minute personalized health education session. Subjects set 3 specific behavior set three specific lifestyle goals prior to discharge including a calculated six month weight loss goal (10% of body weight) and specific dietary and fitness goals. Usual care group participants received no specific instruction regarding weight loss prior to discharge.
  Arms: Intervention Arm
Behavioral: Motivational interviewing and troubleshooting via phone — All subjects were asked to track their weights over the 6 month duration of the study. Weights were obtained by phone at weeks 1,2,3,4, 8, 12, 16, 20 and 24. Phone calls for the intervention group utilized motivational and troubleshooting techniques whereas calls in the usual care group were used only to obtain weight and assess for changes in medications or health condition.
  Arms: Intervention Arm

SUMMARY:
In this study we sought to determine whether inpatient weight loss counseling with post discharge phone follow-up would result in weight loss at six months. Secondary endpoints included weight change from baseline, changes in waist-to-hip ratios, assessment of weight perceptions and changes in patient reported health outcome measures. To our knowledge, this is the first randomized trial designed to evaluate the effects of an obesity intervention with post-discharge follow-up in an inpatient general medicine population.

ELIGIBILITY:
Inclusion Criteria:

* Adults ages 18-65 years old
* Body mass index between 30-50 kg/m2
* Admitted to an internal medicine service

Exclusion Criteria:

* acute medical conditions known to affect weight (heart failure, cirrhosis, end-stage renal disease on dialysis, nephrotic syndrome, or pregnancy)
* Charlson comorbidity index >3
* moderate to severe major depression
* prolonged steroid use (>2 weeks)
* initiation of medications known to affect weight
* non-English speaking
* precontemplation stage of change

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 176 (Actual)
Dates: Start 2011-01; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Weight loss between groups | 6 months

SECONDARY OUTCOMES:
Weight loss from baseline | 6 months
Change in Patient Reported Outcomes Measurement Information System (PROMIS) scores | 6 months
Change in waist-to-hip ratios | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Kelley N Wachsberg, M.D., M.S., Principal Investigator — Northwestern University
Locations (1):
- Northwestern University, Chicago, Illinois, United States